CLINICAL TRIAL: NCT06268353
Title: Is the Plasma Concentration of CAPGDF15 Increased in Pregnancy? A Pilot Study
Acronym: CAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Erik Richter, Professor MD DMSci, University of Copenhagen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 109324-1
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Non-pregnant controls and pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnancy (Experimental): Non-pregnant and pregnant women are compared
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Measure CAPGDF15 in plasma of 3 pregnant and 3 non-pregnant women

SUMMARY:
Background and Purpose During pregnancy, the hormone GDF15 rises between 100-200 times higher than before pregnancy. The significance of this dramatic increase is not clarified, but it has been shown that pregnant women with insufficient increase in GDF15 have a higher risk of spontaneous abortion. CAPGDF15 is a small peptide consisting of 12 amino acids recently found in plasma in both mice and humans, and this peptide is part of the prohormone from which GDF15 is synthesized. Therefore, the assumption is that CAPGDF15 is secreted simultaneously with GDF15. The significance of CAPGDF15 in the organism is completely unknown, except that injection into mice reduces food intake. Therefore, the investigators are interested in investigating whether there is a similar dramatic upregulation of CAPGDF15 as with GDF15 itself. The investigators will not set up a large-scale study without having some prior knowledge of whether this is indeed the case. Therefore, the investigators will conduct a pilot study on 3 pregnant women and 3 control women to examine whether there is any reason to proceed with an actual scientific experiment. Since the increase in GDF15 itself is very large at least100 fold, a pilot study involving only 3 pregnant women and 3 non-pregnant women will be sufficient to gain an impression of whether there is also a significant increase in CAPGDF15. The data will be used to assess whether an actual research project is worth establishing.

Purpose:

The purpose of conducting this pilot study is to investigate whether there is an upregulation of CAPGDF15 similar to that of the hormone GDF15 during pregnancy. By conducting a pilot study on 3 pregnant women and 3 control women, the investigators will see if this is actually the case before setting up an actual scientific experiment.

DETAILED DESCRIPTION:
Experimental Protocol

A total of 6 healthy and fit women will be included in the experiment, 3 pregnant and 3 non-pregnant fertile women matched for age and weight.

Recruitment of Subjects Subjects and matched control subjects will be recruited via Flyers (appendix) posted at the University of Copenhagen.

Inclusion Criteria:

* Healthy and fit pregnant women in the 3rd trimester.
* Healthy control subjects will be matched based on age and weight and must not be taking medication.

Exclusion Criteria:

* Ongoing illness and/or medication intake

Recruitment Procedure and Oral Participant Information The initial contact with a potential participant will be used to address questions about the study. Subsequently, a pre-screening will be conducted over the phone, where inclusion and exclusion criteria will be assessed. Individuals who do not meet the inclusion and exclusion criteria or who do not wish to participate after the initial pre-screening will not be further inconvenienced.

Experimental Day On the 1st and only visit to the experimental site The participant's pregnancy status, gestational week, and age are noted. Weight A routine venous blood sample is taken from one arm vein.

Maximum 1 hour

Outcome Parameters and Method There is no intervention in this experiment. A routine blood sample of 3 ml will be taken from 3 pregnant women and 3 matched non-pregnant control women.

Statistical Considerations:

No formal power calculation has been made, but since the increase in GDF15 itself is significant, 3 pregnant women and 3 non-pregnant women are expected to be sufficient to gain an impression of whether there is also a significant increase in CAPGDF15.

Ethical Considerations:

The project primarily has a basic research perspective. Therefore, there will be no benefits for the participants in participating in the project. The expected basic scientific contribution, in our opinion, will outweigh the discomfort experienced by the participants. Informed consent will be obtained from all participants in accordance with the guidelines of the ethics committee. The experiment, which consists of collecting a single blood sample, will not entail any significant health risks for the participants. If significant information about the participant's health status emerges during the trial period, the participant will be informed, provided consent has been given during the information session. The participant can at any time obtain information about the data - and after the end of the trial information about the result. The trial has been approved by the Ethics Committee RegionH under journal number: Hxxxxxxxx.

Side Effects, Risks, and Disadvantages:

Simple measurements of the body, such as weight and height, are performed using appropriate measuring equipment. These measurements are not expected to entail any risk or discomfort. Blood samples will be taken by the responsible physician. Mild pain may occur at the injection site. In addition, there is a small risk of swelling and tenderness and a small bruise at the injection site, which will disappear after a few days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and fit pregnant women in the 3rd trimester.
* Healthy control subjects will be matched based on age and weight and must not be taking medication.

Exclusion Criteria:

* Ongoing illness and/or medication intake

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
CAPGDF15 levels in plasma | 1 year
  single sample

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - August Krogh Building, Copenhagen
  - University of Copenhagen, August Krogh Section for Molecular Physiology, Copenhagen, Østerbro

IPD SHARING:
Plan to Share IPD: No